CLINICAL TRIAL: NCT03590587
Title: Rapid Structural and Functional Improvements in Following 0.19 mg Fluocinolone Acetonide (FAc) Implant in Diabetic Macular Edema Patients With Poor Visual Acuity: 12-month Audit Results From United Arab Emirates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Collaborators: Sheikh Khalifa Medical City (Other)
Responsible Party: Principal Investigator, Ahmed Elbarky, assistant professor of ophthalmologyu, Benha University
Other Study IDs: skmc
Record Dates: First submitted 2018-07-07; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide; CAF protocol; Drug Implants; Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 1: patients treated with 0.19 mg fluocinolone acetonide (FAc) implant for 12 months
  Interventions: Drug: 0.19 mg fluocinolone acetonide (FAc) implant; Device: 0.19 mg fluocinolone acetonide (FAc) implant

INTERVENTIONS:
Drug: 0.19 mg fluocinolone acetonide (FAc) implant — 0.19 mg fluocinolone acetonide (FAc) implant
Device: 0.19 mg fluocinolone acetonide (FAc) implant — 0.19 mg fluocinolone acetonide (FAc) implant

SUMMARY:
The Health Authority - Abu Dhabi (HAAD) approved the reimbursement of the slow release FAc implant (ILUVIEN) and it is now available for the treatment of diabetic macular edema (DME) in persons who have been previously treated with a course of corticosteroids and did not have a clinically significant rise in intraocular pressure. We performed a retrospective 12-month audit to assess the efficacy and safety of the FAc implant in our clinical practice.

DETAILED DESCRIPTION:
Twenty patients with pseudophakic lenses, treated with ILUVIEN, were investigated to evaluate functional and anatomical characteristics and outcomes (visual acuity [VA; ETDRS letters score], central macular thickness [CMT] and intraocular pressure [IOP]) at baseline, weeks 2-4 and months 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* DME
* Pseudophakic

Exclusion Criteria:

* Other causes of macular edema.
* Phakic
* Know case of gaucoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Twenty patients with pseudophakic lenses, treated with ILUVIEN, were investigated to evaluate functional and anatomical characteristics and outcomes (visual acuity [VA; ETDRS letters score], central macular thickness [CMT] and intraocular pressure [IOP]) at baseline, weeks 2-4 and months 3, 6 and 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-16 (Estimated)

PRIMARY OUTCOMES:
BCVA | 12 months
  best corrected visual acuity

SECONDARY OUTCOMES:
CMT | 12 months
  Central Macular thickness
IOP | 12 months
  Intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Shiekh Khalifa medical city, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided